CLINICAL TRIAL: NCT07040176
Title: Comparison of Distalization of Maxillary First and Second Molars Between a Miniscrew Implant Supported Device and Clear Aligners: A Randomized Clinical Trial.
Brief Title: Comparison of Distalization of Maxillary First and Second Molars Between a Miniscrew Implant Supported Device and Clear Aligners.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Katerina Samandara-Bouzani, Principal investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: protoc.numb. 21/14-12-2023
Record Dates: First submitted 2025-05-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Distalization; Class II Malocclusion; Aligner Therapy; Distalization by Miniscrews
Keywords: Class II malocclusion; Distalization; Orthodontics; Aligners; Miniscrew implants
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AMDA® (Advanced Molar Distalization Appliance) (Active Comparator): The AMDA arm consists of patients that will be treated initially for molar distalization with a miniscrew implant supported device (AMDA®) and for anterior teeth retraction (after molar distalization) with the same device and fixed appliances. The miniscrew implants will be inserted in the anterior region of the palate, especially 6-9 mm posterior to the incisive foramen and 3-6 mm paramedian.
  Interventions: Procedure: Upper molar distalization
- Spark® (Active Comparator): The Spark® arm consists of patients that will be treated with clear aligners and elastics for both molar distalization and anterior teeth retraction.
  Interventions: Procedure: Upper molar distalization

INTERVENTIONS:
Procedure: Upper molar distalization — This study aims to compare upper molar distalization movement achieved with a non-compliance miniscrew implant supported appliance (AMDA®) with distalization of upper molars achieved with clear aligners (Spark®) supported by Class II elastics.

SUMMARY:
The goal of this randomized clinical trial is to compare distalization of maxillary first and second molars achieved with a device supported with mini screw implants in the palate (Advanced Molar Distalization Appliance, AMDA®) with distalization of maxillary first and second molars achieved with clear aligners (Spark®) supported by Class II elastics.

The main questions it aims to answer are:

Is there any difference in achieving upper molar distalization with the Advanced Molar Distalization Appliance (AMDA®) supported by miniscrew implants and with clear aligners (Spark®) supported by Class II elastics at the end of active distalization phase?

Is there any difference between the two groups in the anchorage loss at the end of total treatment?

Additionally, the differences in the movements of premolars, canines and incisors will be analyzed in all three planes of space (sagittal, transverse, vertical), as well as the duration of treatment between the two groups and subgroup comparisons will be performed regarding age, gender, presence of maxillary third molars and severity of malocclusion.

Participants will be randomly assigned to the AMDA® or Spark® group. Treatment will take place at the Department of Orthodontics and participants will have to visit the clinic every 4-6 weeks for regular check ups. Intraoral scans, photographs and x-rays (panoramic x-ray, cephalometric x-rays) will be taken before treatment, at the end of active distalization phase and at the end of treatment.

DETAILED DESCRIPTION:
The aim of the study is to compare distalization of maxillary first and second molars achieved with the Advanced Molar Distalization Appliance (AMDA®) supported by miniscrew implants with distalization of maxillary first and second molars achieved with clear aligners (Spark®) supported by Class II elastics. All patients will be randomly assigned into two groups:

* Group I (AMDA®) consisting of patients that will be treated initially for molar distalization with a miniscrew implant supported device (AMDA®) and for anterior teeth retraction (after molar distalization) with the same device and fixed appliances. The miniscrew implants will be inserted in the anterior region of the palate, especially 6-9 mm posterior to the incisive foramen and 3-6 mm paramedian.
* Group II (Spark®) consisting of patients that will be treated with clear aligners for both molar distalization and anterior teeth retraction.

Lateral cephalometric radiographs of the patients' heads and three-dimensional (3D) intraoral scans of the maxillary and mandibular arches will be taken:

* before treatment (T1),
* at the end of active distalization (T2), (active distalization will be completed, when first and second molars will achieve a full Class I molar relationship (not a super-Class I), and
* at the end of treatment (T3).

Cone Beam Computed Tomography (CBCT) dental scans will be taken in patients assigned to the AMDA group:

* before treatment (T1),
* after miniscrew implant insertion (Tm) CBCT dental scans in T1 will be taken for the 3D evaluation of the anterior palate and the fabrication of a surgical guide for miniscrew implant placement. CBCT dental scans in Tm will verify accuracy of miniscrew implant placement, as well as the existence of enough clearance between miniscrew implants and the roots of upper anterior teeth to ensure a safe retraction of these teeth without the risk of contacting the miniscrew implants and the resulting root resorptions. All CBCT dental scans will be taken in a certified private dental x-ray laboratory.

Completion of orthodontic treatment of all patients will be accomplished when Class I molar and canine relationships, normal overjet and overbite, a good leveling and alignment of the teeth, and a tight occlusion of the posterior teeth will be achieved.

In all these three time points the corresponding 2D and 3D analysis will include:

* angular and linear measurements of the cephalometric analysis,
* angular and linear measurements of the virtual dental casts analysis,
* two-dimensional (2D) superimpositions of the cephalometric tracings, as well as
* 3D superimpositions of the intraoral scans of the maxillary and mandibular arches.
* superimposition of CBCT scans

All patients will be treated in the Postgraduate Clinic of the Department of Orthodontics at the Aristotle University of Thessaloniki by the applicant (Mrs. Samandara) under the supervision of Professor Papadopoulos. Assistance will be provided by the postgraduate students after insertion of the appliance, during the follow up appointments for checking and re-activating the appliances.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least half cusp bilateral Class II malocclusion between upper and lower first molars due to maxillary excess or maxillary protrusion or forward movement of the maxillary posterior teeth, where maxillary molar distalization is indicated.
* Patients in the permanent dentition period of less than 30 years of age with second molars erupted at least one half.
* Patients with good general health and healthy periodontium.

Exclusion Criteria:

* Patients with Class II malocclusion between upper and lower first molars due to mandibular deficiency or mandibular retrusion.
* Patients with less than half cusp bilateral Class II malocclusion between upper and lower first molars.
* Patients with unilateral Class II malocclusion between upper and lower first molars.
* Patients with cleft lip and palate or with other craniofacial syndromes.
* Patients with missing, or congenital missing or supernumerary teeth.
* Patients with full coverage molar restorations.
* Patients with previous orthodontic treatment.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Linear measurements for anteroposterior changes of maxillary first molar distalization movement at the end of active distalization (until Class I molar relationship is achieved). | T1: Baseline records (initial records before the beginning of treatment). T2: 8-12 months, end of distalization phase records (records taken at the end of upper molar distalization, when upper first molars will be bilaterally in Class I malocclusion).
  Cephalometric analysis performed in lateral x-rays and cast analysis performed in intraoral scans will provide us with linear measurements assessing the anteroposterior movement of maxillary first molars.
Linear measurements for anteroposterior changes of maxillary first molar distalization movement at the end of total orthodontic treatment. | T1: Baseline records, (initial records before the beginning of treatment). T3: End of treatment records (records taken at the end of orthodontic treatment after removal of all orthodontic appliances), an average of 24 months.
  Cephalometric analysis performed in lateral x-rays and cast analysis performed in intraoral scans will provide us with linear measurements assessing the anteroposterior movement of maxillary first molars at the end of orthodontic treatment.
Angular measurements for anteroposterior changes of maxillary first molar distalization movement at the end of active distalization (until Class I molar relationship is achieved). | T1: Baseline records (initial records before the beginning of treatment). T2: 8-12 months, end of distalization phase records (records taken at the end of upper molar distalization, when upper first molars will be bilaterally in Class I malocclusion).
  Cephalometric analysis performed in lateral x-rays will provide us with angular measurements assessing the anteroposterior movement of maxillary first molars.
Angular measurements for anteroposterior changes of maxillary first molar distalization movement at the end of total orthodontic treatment. | T1: Baseline records, (initial records before the beginning of treatment). T3: End of treatment records (records taken at the end of orthodontic treatment after removal of all orthodontic appliances), an average of 24 months.
  Cephalometric analysis performed in lateral x-rays will provide us with angular measurements assessing the anteroposterior movement of maxillary first molars at the end of orthodontic treatment.

SECONDARY OUTCOMES:
Duration of active distalization phase | T1: Baseline records (initial records before the beginning of treatment). T2: 8-12 months, at the end of distalization phase (records taken at the end of upper molar distalization, when upper first molars will be bilaterally in Class I malocclusion).
  Comparison of the duration of active distalization between the two approaches (AMDA® and Spark®).
Duration of total treatment | T1: Baseline records, (initial records before the beginning of treatment). T3: End of treatment records (records taken at the end of orthodontic treatment after removal of all orthodontic appliances), an average of 24 months.
  Comparison of the duration of total treatment between the two approaches (AMDA® and Spark®).

CONTACTS AND LOCATIONS:
Overall Officials: Moschos Papadopoulos, Professor, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, School of Medical Sciences, Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD (Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR), Analytic Code will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available 1 month after publication with no end date.
Access Criteria: IPD and supporting information will be shared upon request after contacting the primary investigator of the study.
URL: https://dent.auth.gr/en/postgraduate-program-in-orthodontics-2/

REFERENCES:
- [Background] Wilmes B, Drescher D. Application and effectiveness of the Beneslider: a device to move molars distally. World J Orthod. 2010 Winter;11(4):331-40. PMID 21490998
- [Background] Ravera S, Castroflorio T, Garino F, Daher S, Cugliari G, Deregibus A. Maxillary molar distalization with aligners in adult patients: a multicenter retrospective study. Prog Orthod. 2016;17:12. doi: 10.1186/s40510-016-0126-0. Epub 2016 Apr 18. PMID 27041551
- [Background] Papadopoulos MA, Melkos AB, Athanasiou AE. Noncompliance maxillary molar distalization with the first class appliance: a randomized controlled trial. Am J Orthod Dentofacial Orthop. 2010 May;137(5):586.e1-586.e13; discussion 586-7. doi: 10.1016/j.ajodo.2009.10.033. PMID 20451774
- [Background] Antonarakis GS, Kiliaridis S. Maxillary molar distalization with noncompliance intramaxillary appliances in Class II malocclusion. A systematic review. Angle Orthod. 2008 Nov;78(6):1133-40. doi: 10.2319/101507-406.1. PMID 18947282